CLINICAL TRIAL: NCT03478943
Title: The Real World Study of Apatinib for Gastric Cancer Treatment in Henan Province
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Ahead-HAT01
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators conduct the real world study to explore the efficacy and safety of Apatinib in gastric cancer .

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients .
2. Confirmed by Pathology or histology of Gastric cancer.
3. Patients should be voluntary to the trial and provide with signed informed consent.
4. The researchers believe patients can benefit from the study.

Exclusion Criteria:

1. Patients with a known history of allergic reactions and/or hypersensitivity attributed to apatinib or its accessories.
2. Pregnant or lactating women.
3. Patients with Apatinib contraindications.
4. Patients of doctors considered unsuitable for the trial.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients of gastric cancer in Henan province
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01-30 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Progress free survival | 1 year
Disease-free surviva | 1 year

SECONDARY OUTCOMES:
overall survival | 3 year
Objective Response Rate | 1 year
Disease Control Rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, Principal Investigator — Henan Cancer Hospital; Peichun Sun, Principal Investigator — Henan Provincial People's Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China